CLINICAL TRIAL: NCT02227407
Title: NSC Assistive Technology Research: Reciprocating Gait Orthoses for Paraplegia Patients
Brief Title: Reciprocating Gait Orthoses for Paraplegia Patients
Acronym: UPGO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 201305047RINC; 200703061R (Other: NTUHREC)
Record Dates: First submitted 2014-04-11; First posted 2014-08-28 (Estimated); Last update posted 2014-08-28 (Estimated); Status verified 2014-08

CONDITIONS: Myelomeningocele; Spinal Cord Injury; Spinal Muscular Atrophy
Keywords: SCI; SMA; Paralysis
MeSH Terms: conditions — Meningomyelocele; Spinal Cord Injuries; Muscular Atrophy, Spinal; Paralysis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Energy expenditure, gait pattern, RGOs (Experimental): using motion capture system and forceplates to monitor gait pattern while wearing reciprocating gait orthoses to calculate the mechanical energy cost
  Interventions: Device: RGOs(reciprocating gait orthoses)

INTERVENTIONS:
Device: RGOs(reciprocating gait orthoses) — using additional apparatus combined with Hip-Knee-Ankle-Foot orthoses (HKAFO) to help paraplegia patients to present reciprocating gait pattern
  Other Names: other name:HKAFO(Hip-Knee-Ankle-Foot orthoses)

SUMMARY:
Ambulation would bring many physiological and psychological benefits and getting up and walking has been a dream for paraplegia patients.The reciprocating gait orthoses (RGOs) for paraplegics particularly draws research attentions because it mimics human gait pattern.But, the high energy consumption and low walking speeds caused the frequent abandonment or the low utilization of the reciprocating gait orthoses.To improve the design reducing the energy expenditure, it requires biomechanical analysis of the pathological gait such that the gait deviations and energy consuming mechanisms can be identified and remedial means can be implemented.

The investigators hypotheses will include that there would exist an energy saving mechanism of human reciprocating locomotion based on the principle of conservation of mechanical energy.Secondly, kinematic and kinetic gait determinants could be derived from the energy saving mechanism. Finally, the control of knee joint coordinating with the hip joint movements would facilitate the gait progression and further reduce the energy consumption.

The objective of this clinical trial is to evaluate the gait of paraplegic patients with reciprocating gait orthoses and to support the investigators research in biomechanical analysis, design and control of reciprocating gait orthoses for paraplegia patients. An experiment to study the pathological gait of paraplegia patients with an existing reciprocating gait orthosis will be carried out.

DETAILED DESCRIPTION:
Background: Ambulation is a rehabilitation priority for many paraplegic patients, either for the psychological reasons or with the aim to achieve partial or full independence. It also provides the therapeutic benefits which are widely acknowledged to improve urinary drainage, to improve peripheral circulation, and to prevent the complication caused from bedridden, such as contracture, osteoporosis, urinary tract infection, and constipation etc. Some studies also found that ambulation will increase cardiopulmonary function. For those pediatric spinal cord-injured patients, the upright posture also profits the development of trunk and head control. There are a number of reciprocating gait orthoses (RGOs) available in practice for paraplegics, the problems of which have been slow, heavy and high energy-consumption. The biomechanical causes are not fully understood. Despite all the benefits that RGOs can offer, research and clinical experience indicated that most paraplegia patients choose wheelchair mobility after discharge to the community because it is faster, safer and needs less energy expenditure. Therefore, a biomechanical study of the pathological gait of paraplegia patients with RGOs is critically needed. The problems of currently applied RGOs need to be analyzed and remedial means to be proposed. In addition, a new RGOs system is also needed to serve as a research tool and a platform proving the remedial ideas.

Literature Review: There are many kinds of gait orthoses prescribed for paraplegics, which can be grouped according to the patterns of propulsion. The first type is a group of swing-through gait orthoses which include the Knee-Ankle-Foot orthoses (KAFO), Hip-Knee-Ankle-Foot orthoses (HKAFO), and the parapodium. The swing-through gait has high energy cost and users give up the orthoses easily. Swivel walkers belong to the second group, which enables paraplegic patients to ambulate in an upright position without the use of crutches or other walking aids. Patients progress by shifting the center of gravity; and increase the walking speed by swing their arms and by the rotation of the trunk. Loretta et al. compared the swivel gait with the swing gait, which shows the swivel gait has slower speed but more efficient gait which implies that lower metabolic cost and oxygen consumption are needed. Although the swivel walker has the advantages of providing low energy and hand-free walking, it was most criticized for its low walking speed and for its inability to ambulate on an uneven surface. The third one is a group of reciprocating gait orthoses which were developed with a belief that they would provide a more energy efficient gait than other gait orthoses. The LSU RGOs developed in the early 1980's has hip joints that are linked to act in a reciprocal pattern. In the early 1990s, there were two revised version of the LSU RGOs developed, ARGOs (Advanced RGOs using one cable and IRGOs (Isocentric RGOs) using a solid rocker bar. The hip guidance orthosis (HGOs) that provides friction-free hip joint also allows patients to walk reciprocally. WO, walkabout orthosis, is an infraperineal structure that also facilitates reciprocating walking. Comparing with HKAFO, RGOs was heavier, slower, and the energy cost (mL/kg/m) was higher although the energy consumption rate (mL/kg/min) was significantly higher for children in HKAFOs.

To achieve an efficient gait and to overcome the problem to be slow, the hybrid system, that is the combination of the FES and RGOs , had shown the possibility for improvement. Because this system used both the RGOs structural stability and muscle power stimulated by FES to decrease the activity of the trunk muscles in prevention from fatigue, it can provide more energy-efficient gait that increases the aerobic-anaerobic threshold of the patients in the long term.

Many orthotic options for paraplegia are available but only to provide limited walking functions with great energy consumption, which has been the reason for the frequent abandonment or the low utilization of the RGOs. To improve the design reducing the energy expenditure, it requires biomechanical analysis of the pathological gait such that the gait deviations and energy consuming mechanisms can be identified and remedial means can be implemented. There has been a recent research on the biomechanical analysis of an ARGOs user's gait and some possible mechanisms contributing to the high energy consumption were discussed. However, no further remedial action in terms of design parameters was suggested in their work. It is obvious that more research on the biomechanical study are needed to advance the development of orthotic solutions for paraplegia patients.

Gait determinants were to identify the sources which affect the energy expenditure. The determinants include pelvic rotation, pelvic list, knee flexion at mid-stance, foot and ankle motion, knee motion and lateral pelvic displacement. There were studies to evaluate the effects of these kinematic gait determinants on reduction of the vertical displacement of the Body Center of mass (BCOM). Gard and Childress found that the magnitude of the trunk's vertical excursion was virtually unaffected by pelvic list. Kerrigan pointed out the there are other primary gait determinants needed to explain the actual reduction in BCOM vertical displacement. A reduction of BCOM vertical excursion may have significant energy implications, but it requires kinetic consideration to prove the gait determinants do affect the energy expenditure.

Kinetic consideration was given in studies to the analysis of mechanical energy emphasizing the exchange between potential and kinetic energy. A study of normal subjects suggested a greater exchange between potential and kinetic energy near individually preferred walking speeds. Since it was previously found that the self-selected speed minimizes the energy cost, it can be readily induced that the normal gait with lower energy cost implies a greater conservation of mechanical energy, i.e., a greater exchange between potential and kinetic energy. It remains unclear as to what roles the gait determinants play in conserving the mechanical energy.

In addition, joint biomechanics in the dynamic coordination particularly could never be overemphasized when the energy consumption during ambulation is concerned. Gait efficiency in terms of energy cost for ankle fusion patients reached 90% but the hip fusion patients achieved only a 53% gait efficiency. The ankle fusion does not require major compensatory movements in the gait pattern but only local substitutions in mid and forefoot areas were observed. When the hip and the knee were disturbed, patients require pay in energy consumption and compensatory substitutions for the lost function in the hip and the knee. It implies that coordination of the knee and the hip has higher priority than the ankle and human coordinating knee and hip movements could negotiate fairly well even with ankle disturbance in walking to maintain energy consumption and speeds.

A hybrid orthosis system (HOS) has been being studied for walking after spinal-cord injury (SCI), which coordinates the mechanical locking and unlocking of knee and ankle joints of a reciprocating gait orthoses, while propulsive forces are injected and unlocked joints controlled with functional neuromuscular stimulation. A feasibility study was carried out for a functional neuromuscular stimulation powered mechanical gait orthosis with coordinated joint locking (stance control KAFO). A laboratory hybrid RGOs was developed using a HKAFO which contains controllable friction brakes at both hip and knee joints. A computer-controlled orthosis system has been developed to address the problems of rapid muscle fatigue and poor movement control that are characteristic of FES-aided gait. However, the theme was not on the hip and knee coordination. In order that the coordination of hip and knee joints can be studied, a computer simulation and experiment validation are necessary. Therefore, a research tool needs to be developed so that a study can be conducted on the effectiveness of the knee and hip coordination on the reduction of energy expenditure during ambulation in paraplegia patients with reciprocating gait orthoses.

Research Objectives: In this research, the investigators hypotheses will include that there would exist an energy saving mechanism of human reciprocating locomotion based on the principle of conservation of mechanical energy.Secondly, kinematic and kinetic gait determinants could be derived from the energy saving mechanism. Finally, the control of knee joint coordinating with the hip joint movements would facilitate the gait progression and further reduce the energy consumption.

Experimental equipments, devices and protocols: The patient evaluation, RGOs design and fabrication, and fitting will be done under supervision of qualified orthotists in the Rehabilitation Engineering Research Center at National Taiwan University (NTURERC). A Cosmed K4b2 portable gas analysis system will be used to acquire physiological measures such as heart rates and oxygen consumption. A three dimensional motion measurement system (Optotrak® Certus™, Northern Digital Inc., Waterloo, Ontario, Canada) with two position sensors, each with three cameras, will be used to collect kinematic data. Twelve rigid bodies with active markers will be attached on the segments of subjects of the left upper arms, thighs, shanks, heels, and the pelvis and the trunk. Eight force plates (AMTI) will be used to calculate the kinetics of the segments of the lower limbs when using assistance. Participants will be given instructions for the experiment. Patient's medical data such as diagnosis, onset, birth date, gender, height and weight will be taken and basic data of normal subjects' will be collected as well. Paraplegic subjects will walk at their self selected speeds and complete at least three trials. The kinematic and kinetic data will be collected synchronously. Patients will be asked to walk at their self selected speed for 30 meters along a designated route three times in order to measure heart rates and oxygen consumption.

ELIGIBILITY:
Inclusion Criteria:

* myelomeningocele or spinal cord injured patients at neurological level of T10-L2).
* they should be walking with RGO for at least 30 meters (assistant device if needed).

Exclusion Criteria:

* spasticity, contractures, and recurrent lower limb injuries
* other neuromuscular disease
* insufficient walking ability

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2013-08; Primary Completion 2015-12 (Estimated); Study Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
the difference of joint kinetic data in able-bodied subjects and RGO users | baseline, 30 minutes after fitting of the RGOs
  joint force, joint moment and joint power during gait

SECONDARY OUTCOMES:
the difference of gait parameter in able-bodied subjects and RGO users | baseline, 30 minutes after fitting of the RGOs
  stride length, gait cycle period, gait speed
the difference of joint kinematic data in able-bodies subjects and RGO users | baseline, 30 minutes after fitting of the RGOs
  joint angle, joint excursion, joint angular velocity and acceleration

OTHER OUTCOMES:
the difference of energy flow in able-bodied subjects and RGO users | baseline, 30 minutes after fitting of the RGOs
  measurement of the joint and segmental mechanical energy transfer during gait while using orthoses

CONTACTS AND LOCATIONS:
Overall Officials: Liang-Wey Chang, Ph.D., Principal Investigator — Rehabilitation Engineering Lab,NTU
Locations (1):
- Rehabilitation Engineering Research Center, Taipei, Taiwan, Taiwan